CLINICAL TRIAL: NCT00330642
Title: Rapid Detection of Group B Streptococcus Using a Bedside Microfluidics Device: Labor and Delivery Study
Brief Title: Rapid Detection of Group B Streptococcus (Strep)-Labor and Delivery Study
Status: Withdrawn | Type: Observational
Why Stopped: HandyLab device did not work for the science
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mark Pearlman, S Jan Behrman Collegiate Professor of Reproductive Medicine, Professor of Obstetrics and Gynecology and Professor of Surgery, Medical School, University of Michigan
Other Study IDs: HandyLab #VVP00103
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Streptococcal Infections
Keywords: Streptococcus Group B; Pregnancy
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether a rapid bedside diagnosis of group B strep (GBS) growing in the vagina and rectum can be performed with similar success to the routine culture in women who are in labor.

DETAILED DESCRIPTION:
Group B Strep neonatal infections is one of the leading infections in newborns, most of which are acquired by vertical transmission at the time of childbirth. Most cases can be prevented by identifying women who are colonized with GBS in the vaginal-rectal area and giving colonized women prophylactic antibiotics in labor. About 15-20% of women are colonized and nearly all of these women are asymptomatic. Because it takes up to 48 hours to obtain culture results, it is currently recommended to perform cultures in the clinic about 5 weeks prior to their due date and then treat those with GBS when they come in for labor. There are several downsides to this strategy. All women who present with preterm labor are treated until culture results become available (overtreatment); women who go into labor while waiting for culture results are all treated (overtreatment); prior studies have shown 33% of women are positive at 35 weeks, but negative at birth (overtreatment) and 10% are negative at 35 weeks and positive at birth (undertreatment); lost or missing culture results (over- or undertreatment). Using microfluidics and fluorescent PCR, a new test can identify GBS reliably in 30 to 45 minutes in vitro. This study proposes to evaluate the clinical performance (sensitivity, specificity, positive and negative predictive value) of the microfluidic rapid GBS technique in un-selected sequential women presenting to labor and delivery, comparing them to cultures taken at the same time and the 35-37 week cultures in these same women. We will also evaluate the identification of GBS before and after rupture of membranes (amniotomy) using both standard GBS culture and rapid PCR (HandyLab technology).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Mentally capable of giving informed consent
* Symptoms and signs at presentation related to possible labor or ruptured membranes (leakage of fluid, uterine contractions, pelvic pressure)
* Presentation for induction of labor irrespective of cause

Exclusion Criteria:

* Inability to give informed consent
* Conditions where the time taken to obtain specimens are potentially harmful to one or one's baby (heavy bleeding, low fetal heart rate, preterm premature rupture of membranes)
* Use of any antibacterials within the previous 7 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older who present for induction of labor.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pearlman, MD, Principal Investigator — University of Michigan, Obstetrics and Gynecology
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Boyer KM, Gotoff SP. Prevention of early-onset neonatal group B streptococcal disease with selective intrapartum chemoprophylaxis. N Engl J Med. 1986 Jun 26;314(26):1665-9. doi: 10.1056/NEJM198606263142603. PMID 3520319
- [Background] Yancey MK, Schuchat A, Brown LK, Ventura VL, Markenson GR. The accuracy of late antenatal screening cultures in predicting genital group B streptococcal colonization at delivery. Obstet Gynecol. 1996 Nov;88(5):811-5. doi: 10.1016/0029-7844(96)00320-1. PMID 8885919
- [Background] Schrag S, Gorwitz R, Fultz-Butts K, Schuchat A. Prevention of perinatal group B streptococcal disease. Revised guidelines from CDC. MMWR Recomm Rep. 2002 Aug 16;51(RR-11):1-22. PMID 12211284
- [Background] Edwards RK, Clark P, Duff P. Intrapartum antibiotic prophylaxis 2: positive predictive value of antenatal group B streptococci cultures and antibiotic susceptibility of clinical isolates. Obstet Gynecol. 2002 Sep;100(3):540-4. doi: 10.1016/s0029-7844(02)02097-5. PMID 12220775
- [Background] ACOG committee opinion. Prevention of early-onset group B streptococcal disease in newborns. Number 173--June 1996. Committee on Obstetric Practice. American College of Obstetrics and Gynecologists. Int J Gynaecol Obstet. 1996 Aug;54(2):197-205. No abstract available. PMID 9236325
- [Background] Centers for Disease Control and Prevention (CDC). Laboratory practices for prenatal Group B streptococcal screening and reporting--Connecticut, Georgia, and Minnesota, 1997-1998. MMWR Morb Mortal Wkly Rep. 1999 May 28;48(20):426-8. PMID 10365633
- [Background] Yancey MK, Armer T, Clark P, Duff P. Assessment of rapid identification tests for genital carriage of group B streptococci. Obstet Gynecol. 1992 Dec;80(6):1038-47. PMID 1448249
- [Background] Walker CK, Crombleholme WR, Ohm-Smith MJ, Sweet RL. Comparison of rapid tests for detection of group B streptococcal colonization. Am J Perinatol. 1992 Jul;9(4):304-8. doi: 10.1055/s-2007-999247. PMID 1627226
- [Background] Bergeron MG, Ke D, Menard C, Picard FJ, Gagnon M, Bernier M, Ouellette M, Roy PH, Marcoux S, Fraser WD. Rapid detection of group B streptococci in pregnant women at delivery. N Engl J Med. 2000 Jul 20;343(3):175-9. doi: 10.1056/NEJM200007203430303. PMID 10900276